CLINICAL TRIAL: NCT01332968
Title: A Multicenter, Phase III, Open-Label, Randomized Study in Previously Untreated Patients With Advanced Indolent Non-Hodgkin's Lymphoma Evaluating the Benefit of GA101 (RO5072759) Plus Chemotherapy Compared With Rituximab Plus Chemotherapy Followed by GA101 or Rituximab Maintenance Therapy in Responders
Brief Title: A Study of Obinutuzumab (RO5072759) Plus Chemotherapy in Comparison With Rituximab Plus Chemotherapy Followed by Obinutuzumab or Rituximab Maintenance in Patients With Untreated Advanced Indolent Non-Hodgkin's Lymphoma (GALLIUM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: German Low Grade Lymphoma Study Group (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21223; 2010-024132-41 (EudraCT Number)
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — obinutuzumab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Bendamustine Hydrochloride; Rituximab

ARMS (2):
- Rituximab+Chemotherapy (Active Comparator): Participants will receive either 8 cycles of rituximab along with 6 cycles of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) (21-day cycle) or 8 cycles of rituximab along with 8 cycles of cyclophosphamide, vincristine, and prednisone (CVP) (21-day cycles) or 6 cycles of rituximab along with 6 cycles of bendamustine (28-day cycle) during the induction period. The induction period will be followed by either a maintenance or observation period for responders or non-responders, respectively. Responders will receive rituximab monotherapy every 2 months for 2 years during the maintenance period. Non-responders will receive no protocol specified treatment during the 2-year observation period. Finally, participants will be followed during a 5-year follow-up period. The chemotherapy regimen (CHOP or CVP or bendamustine) for individual participant will be chosen by the site prior to initiation of the study.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Bendamustine; Drug: Rituximab
- Obinutuzumab+Chemotherapy (Experimental): Participants will receive either 8 cycles of obinutuzumab along with 6 cycles of CHOP (21-day cycle) or 8 cycles of obinutuzumab along with 8 cycles of CVP (21-day cycles) or 6 cycles of obinutuzumab along with 6 cycles of bendamustine (28-day cycle) during induction period. The induction period will be followed by either a maintenance or observation period for responders or non-responders, respectively. Responders will receive obinutuzumab monotherapy every 2 months for 2 years during the maintenance period. Non-responders will receive no protocol specified treatment during the 2-year observation period. Finally, participants will be followed during a 5-year follow-up period. The chemotherapy regimen (CHOP or CVP or bendamustine) for individual participant will be chosen by the site prior to initiation of the study.
  Interventions: Drug: Obinutuzumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Bendamustine

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab 1000 milligrams (mg) intravenous (IV) infusion will be administered on Day 1, 8, and 15 of Cycle 1 and then on Day 1 of each subsequent cycle during induction period and obinutuzumab 1000 mg IV infusion every 2 months during maintenance period.
  Other Names: GA101; RO5072759
  Arms: Obinutuzumab+Chemotherapy
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m^2 IV will be administered on Day 1 of each cycle during induction period.
Drug: Doxorubicin — Doxorubicin 50 mg/m^2 IV will be administered on Day 1 of each cycle during induction period.
Drug: Vincristine — Vincristine 1.4 mg/m^2 (maximum 2 mg) IV will be administered on Day 1 of each cycle during induction period.
Drug: Prednisone — Prednisone 100 mg (or equivalent prednisolone or methylprednisolone) will be administered orally on Days 1-5 of each cycle during induction period.
Drug: Bendamustine — Bendamustine 90 mg/m^2 IV infusion will be administered on Days 1 and 2 of each cycle during induction period.
Drug: Rituximab — Rituximab 375 milligrams per square meter (mg/m^2) IV infusion will be administered on Day 1 of each cycle during induction period and rituximab 375 mg/m^2 every 2 months during maintenance period.
  Other Names: MabThera/Rituxan
  Arms: Rituximab+Chemotherapy

SUMMARY:
This open-label, randomized study will assess the efficacy and safety of obinutuzumab (RO5072759) in combination with chemotherapy compared to rituximab (MabThera/Rituxan) with chemotherapy followed by obinutuzumab or rituximab maintenance in participants with untreated advanced indolent non-Hodgkin's lymphoma. After the end of the induction period, participants achieving response (Complete response [CR] or partial response [PR]) will undergo a maintenance period continuing on the randomized antibody treatment alone every 2 months until disease progression for a total of 2 years. Anticipated time on study treatment is up to approximately 2.5 years. After maintenance or observation, participants will be followed for 5 years until progression. After progression, participants will be followed for new anti-lymphoma therapy and overall survival until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Cluster of differentiation 20 (CD20)-positive indolent B-cell non-Hodgkin's lymphoma (follicular lymphoma or splenic, nodal or extranodal marginal zone lymphoma)
* Stage III or IV disease, or Stage II bulky disease (defined as tumor diameter greater than or equal to [>/=] 7 centimeters [cm])
* For participants with follicular lymphoma: requirement for treatment according to Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria
* For participants with symptomatic splenic, nodal, or non-gastric extranodal marginal zone lymphoma: disease that is de novo or has relapsed following local therapy (i.e. surgery or radiotherapy) and requires therapy as assessed by the investigator
* At least one bi-dimensionally measurable lesion (greater than [>] 2 cm in its largest dimension by computed tomography [CT] scan or magnetic resonance imaging [MRI])
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Adequate hematologic function

Exclusion Criteria:

* Central nervous system lymphoma, leptomeningeal lymphoma, or histological evidence of transformation to a high-grade or diffuse large B-cell lymphoma
* Grade 3b follicular lymphoma, small lymphocytic lymphoma or Waldenström's macroglobulinaemia
* Ann Arbor Stage I disease
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Known hypersensitivity to any of the study drugs or sensitivity to murine products, or history of sensitivity to mannitol
* For participants with follicular lymphoma: prior treatment for non-Hodgkin's lymphoma with chemotherapy, immunotherapy, or radiotherapy
* For participants with non-follicular lymphoma: prior treatment with chemotherapy or immunotherapy
* Regular treatment with corticosteroids during the 4 weeks prior to the start of Cycle 1
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results
* For participants who will be receiving cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP): left ventricular ejection fraction (LVEF) less than (<) 50% by multiple-gated acquisition (MUGA) scan or echocardiogram
* History of prior other malignancy with the exception of curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix at any time prior to study
* Known active infection, or major episode of infection within 4 week prior to the start of Cycle 1
* Vaccination with a live vaccine within 28 days prior to randomization
* Recent major surgery (within 4 weeks prior to start of Cycle 1), other than for diagnosis
* Abnormal laboratory values as defined by protocol for creatinine, creatinine clearance, aspartate transaminase (AST) or alanine transaminase (ALT), total bilirubin, international normalized ration (INR), partial thromboplastin time (PTT) or activated partial thromboplastin time (aPPT), unless these abnormalities are due to underlying lymphoma
* Positive test results for human immunodeficiency virus (HIV), human T-lymphotropic virus 1 (HTLV1), hepatitis C or chronic hepatitis B
* Pregnant or lactating women
* Life expectancy <12 months
* Participation in another clinical trial with drug intervention within 28 days prior to start of Cycle 1 and during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1401 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (183):
- United States (12):
  - Highlands Oncology Group, Springdale, Arkansas
  - The Regents of the University of California; Office of Research, Irvine, California
  - Kootenai Cancer Center, Post Falls, Idaho
  - Illinois Cancer Care, P.C. - Galesburg, Galesburg, Illinois
  - Siouxland Hematology/Oncology, Sioux City, Iowa
  - University of Kansas; Medical Center & Medical pavilion, Westwood, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Mercy Medical Research Institute, Springfield, Missouri
  - MT Cancer Inst Fndtn; MT Can Spec, Missoula, Montana
  - San Juan Oncology Associates, Farmington, New Mexico
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (8):
  - Concord Repatriation General Hospital; Haematology, Sydney, New South Wales
  - Westmead Hospital; Haematology, Sydney, New South Wales
  - Princess Alexandra Hospital Woolloongabba; Clinical Hematology and Medical Oncology, Woolloongabba, Queensland
  - St Vincent'S Hospital; Haematology, Fitzroy, Victoria
  - Peter MacCallum Cancer Centre; Department of Haematology, Melbourne, Victoria
  - Austin and Repatriation Medical Centre; Cancer Services, Melbourne, Victoria
  - Monash Medical Centre; Haematology, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (3):
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
- Canada (8):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Dr. Georges L. Dumont University Hospital Centre, Moncton, New Brunswick
  - Ottawa General Hospital, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Toronto East General Hospital; Haematology/Oncology, Toronto, Ontario
  - Hopital Charles Lemoyne; Centre Integre de Lutte Contre Le Cancer de La Monteregie, Greenfield Park, Quebec
- China (13):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Peking University First Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - General Hospital of Chinese PLA; Department of Hematology, Beijing
  - the First Hospital of Jilin University, Changchun
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Province Hospital, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Union Hospital of Tongji Medical College, Dept. of Cancer Center; Cancer Center, Wuhan
- Czechia (3):
  - Fakultni nemocnice Brno; Interni hematologicka a onkologicka klinika, Brno
  - Fn Hr. Kralove; IV. Interni Hematologicka Klinika, Hradec Králové
  - Vseobecna Fakultni Nemocnice v Praze, I. Interni Klinika - Klinika Hematoonkologie VFN a 1. LF UK, Prague
- Helsinki University Central Hospital; Dept of Oncology, Helsinki, Finland
- France (7):
  - Hotel Dieu; Medecine D, Angers
  - Hopital Augustin Morvan; Hematologie, Brest
  - Chu Estaing; Hematologie Clinique Adultes, Clermont-Ferrand
  - Clinique Victor Hugo, LeMans
  - Hopital De La Conception; Hematologie Clinique, Marseille
  - Hopital Saint Eloi; Hematologie Oncologie Medicale, Montpellier
  - Hopital Saint Jean; Hematologie, Perpignan
- Germany (45):
  - Onkologischer Schwerpunkt am Oskar-Helene-Heim; Dres. Herrenberger, Keitel-Wittig u. Kirsch, Berlin
  - Klinikum Chemnitz gGmbH Krankenhaus Küchwald Klinik f.Innere Medizin III, Chemnitz
  - Klinik der Uni zu Köln; Klinik für Innere Medizin, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Gemeinschaftspraxis Dr. med. J. Mohm und Dr. med. G. Prange-Krex; Fachaerzte fuer Innere Medizin, Dresden
  - HELIOS Klinikum Erfurt I.Medizinische Klinik, Erfurt
  - St.-Antonius-Hospital gGmbH; Klinik für Hämatologie und Onkologie, Eschweiler
  - Universitätsklinikum Essen; Innere Klinik und Poliklinik für Tumorforschung, Essen
  - Klinik Johann Wolfgang von Goethe Uni; Medizinische Klinik II, Frankfurt
  - Universitätsklinikum Freiburg; Klinik für Innere Medizin I; Hämatologie/Onkologie, Freiburg im Breisgau
  - Uni Göttingen, Georg-August-Universität; Klinik für Hämatologie und Medizinische Onkologie, Göttingen
  - Universitätsklinikum Greifswald Klinik für Innere Medizin C und Poliklinik, Greifswald
  - Kath. Krankenhaus Hagen gem. GmbH, St.-Josefs-Hospital; Klinik für Hämatologie und Onkologie, Hagen
  - Onkologische Schwerpunktpraxis Dres. Bernd Gaede, Hans-Ulrich Ehlers, Ulrike Rodewig u.w., Hanover
  - Dres.Andreas Karcher und Stefan Fuxius, Heidelberg
  - Uniklinik Heidelberg, Medizinische Klinik & Poliklinik V, Heidelberg
  - Universitaetsklinikum des Saarlandes; medizinische Klinik und Poliklinik; Innere Medizin I, Homburg/Saar
  - Universitätsklinikum Jena; Klinik für Innere Medizin II, Jena
  - UKSH, Campus Kiel; Klinik für Innere Medizin II, Hämatologie und Internistische Onkologie, Kiel
  - Institut für Versorgungsforschung in der Onkologie GbR Koblenz, Koblenz
  - Tagesklinik Landshut; Hämatologie/Onkologie, Landshut
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Lebach
  - Klinikum St.Georg gGmbH Klinik für Internistische Onkologie und Hämotologie, Leipzig
  - Klinikum der Stadt Ludwigshafen; Medizinische Klinik A, Ludwigshafen
  - Onkologische Gemeinschaftspraxis, Magdeburg
  - Otto von Guericke Uni Magdeburg Uniklinik; Hämatologie/Onkologie, Magdeburg
  - Uni. der Johannes Gutenberg-Universitaet Mainz; III. Medizinische Klinik und Poliklinik, Mainz
  - Mannheimer Onkologie Praxis Dres. Jürgen Brust Dieter Schuster, Mannheim
  - Klinikum Mannheim III. Medizinische Klinik, Mannheim
  - St. Frankziskus Krankenhaus, Med. Klinik I; Klinik für Hämatologie,Onkologie u. Gastroenterologie, Mönchengladbach
  - Kliniken Ostalb, Stauferklinikum Schwäbisch-Gmünd; Zentrum für Innere Medizin, Mutlangen
  - Klinikum der Universität München, Campus Großhadern; Medizinische Klinik und Poliklinik III, München
  - Klinikum rechts der Isar der TU München; III. Medizinischen Klinik (Hämatologie/Onkologie), München
  - Gemeinschaftspraxis Dr. med. Holger Klaproth, Neunkirchen/Saar
  - Pius-Hospital; Klinik fuer Haematologie und Onkologie, Oldenburg
  - Brüderkrankenhaus St. Josef, Paderborn
  - Prosper-Hospital, Medizinische Klinik I, Recklinghausen
  - Krankenhaus Barmherziger Brüder; Klinik für Internistische Onkologie / Hämatologie, Regensburg
  - Praxis für Hämatologie & Onkologie, Saarbrücken
  - Krankenhaus der Barmherzigen Brüder Trier; Innere Medizin I, Hämatologie / Internistische Onkologie, Trier
  - Universität Tübingen; Med. Klinik; Innere Medizin I, Tübingen
  - Universtitätsklinikum Ulm; Klinik für Innere Medizin III, Ulm
  - Helios Dr. Horst Schmidt Kliniken; Klinik Innere MED III: Hämatologie, Onkologie, Palliativmedizin, Wiesbaden
  - Hämatologisch-Onkologische Schwerpunktpraxis Dres. Schlag & Schöttker, Würzburg
- Hungary (5):
  - Semmelweis University, First Dept of Medicine, Budapest
  - National Institute of Oncology, A Dept of Internal Medicine, Budapest
  - University of Debrecen Medical and Health Science Center, Institute of Internal Medicine, Hematology, Debrecen
  - Petz Aladar Megyei Korhaz; Hematologia, Győr
  - University of Szeged, II Dept of Internal Medicine, Szeged
- Israel (3):
  - Rambam Medical Center; Heamatology & Bone Marrow Transplantation, Haifa
  - Beilinson Medical Center; Haematology, Petah Tikva
  - Chaim Sheba Medical Center; Hematology BMT & CBB, Ramat Gan
- Italy (9):
  - Azienda Ospedaliera Universitaria di Modena, Modena, Emilia-Romagna
  - Az. Osp. S. Camillo Forlanini; Uo Ematologia E Trapianti Di Midollo Osseo, Rome, Lazio
  - ASST PAPA GIOVANNI XXIII; Ematologia, Bergamo, Lombardy
  - Ospedale Maggiore Di Milano; U.O. Ematologia I - Padiglione Marcora, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Istituto Clinico Humanitas;U.O. Oncologia Medica Ed Ematologia, Rozzano, Lombardy
  - Ospedale V. Cervello; U.O. Ematologia E Trapianti, Palermo, Sicily
  - A.O. Univ.Ospedali Riuniti Umerto I -G.M.Lancisi G.Salesi; U.O. Clinica Di Ematologia, Torrette DI Ancona, The Marches
  - Uni Degli Studi; Dip.Med.Clinica E Sperim. Ematologia, Padua, Veneto
- Japan (24):
  - Aichi Cancer Center Hospital; Hematology and Cell Therapy, Aichi
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital; Hematology & Oncology, Aichi
  - Nagoya City University Hospital; Hematology and Oncology, Aichi
  - Aomori Prefectural Central Hospital; Hematology, Aomori
  - Chiba Cancer Center;Hematology and Oncology, Chiba
  - National Cancer Center Hospital East;Hematology, Chiba
  - Shikoku Cancer Center; Hematology and Oncology, Ehime
  - National Hospital Organization Kyushu Cancer Center; Hematology, Fukuoka
  - Gunma University Hospital;Hematology, Gunma
  - Hiroshima University Hospital; Hematology, Hiroshima
  - Kobe City Medical Center General Hospital; Hematology, Hyōgo
  - Hyogo Cancer Center; Department of hematology, Hyōgo
  - Tokai University Hospital; Hematology, Kanagawa
  - Kumamoto University Hospital; Hematology Rheumatology and Clinical Immunology, Kumamoto
  - University Hospital, Kyoto Prefectural University of Medicine; Hematology, Kyoto
  - Tohoku University Hospital; Hematology and Immunology, Miyagi
  - Shinshu University Hospital; Hematology, Nagano
  - Niigata Cancer Center Hospital; Internal Medicine, Niigata
  - Matsushita Memorial Hospital; hematology, Osaka
  - Jichi Medical University Hospital; Hematology, Tochigi
  - National Cancer Center Hospital; Hematology, Tokyo
  - Toranomon Hospital; Hematology, Tokyo
  - The Cancer Institute Hospital of JFCR; Hematology Oncology, Tokyo
  - The Jikei University Daisan Hospital; Department of Clinical Oncology and Hematology, Tokyo
- Russia (3):
  - FSBI Russian Oncology Research Center n.a. Blokhin of MOH RF, Moscow
  - Regional Clinical Hospital N.A. Semashko; Hematology, Nizhny Novgorod
  - Republican Clinical Hospital n.a. Baranov; Haematology, Petrozavodsk
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol; Servicio de Hematologia, Badalona, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Hematologia, Sabadell, Barcelona
  - Fundacion Hospital de Alcorcon; Servicio de Hematologia, Alcorcón, Madrid
  - Hospital de Basurto; Servicio de Hematologia, Bilbao, Vizcaya
  - Hospital Univ. 12 de Octubre; Servicio de Hematologia, Madrid
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
- Sahlgrenska Universitetssjukhuset; Sektionen för hematologi och koagulation, Gothenburg, Sweden
- Taiwan (3):
  - National Taiwan Universtiy Hospital; Division of Hematology, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
  - Chang Gung Medical Foundation - Linkou; Division of Hematology- Oncology, Taoyuan District
- United Kingdom (29):
  - Aberdeen Royal Infirmary; Haematology - Ward 16, Aberdeen
  - Queen Elizabeth Hospital; Centre for Clinical Haematology, Birmingham
  - Royal Bournemouth General Hospital; Haematology, Bournemouth
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrookes Hospital; Haematology, Cambridge
  - Kent & Canterbury Hospital; Clinical Haematology, Canterbury
  - Velindre NHS Trust; Haematology Department, Cardiff
  - Castle Hill Hospital; The Queens Centre for Oncology and Haematology, Cottingham
  - Western General Hospital; Department of Haematology, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - James Paget Hospital; Haematology Department, Great Yarmouth
  - Princess Alexandra Hospital; Department of Haematology, Harlow
  - St James Uni Hospital; Icrf Cancer Medicine Research Unit, Leeds
  - Leicester Royal Infirmary; Dept of Haematology, Leicester
  - St Bartholomew's Hospital, London
  - King'S College Hospital; Haematology, London
  - St. George'S Hospital; Haematology, London
  - Hammersmith Hospital; Haematology, London
  - University College Hospital; Macmillan Cancer Centre, London
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Norfolk & Norwich Hospital; Dept of Haematology, Norwich
  - Nottingham City Hospital; Dept of Haematology, Nottingham
  - Churchill Hospital; Oxford Cancer and Haematology Centre, Oxford
  - Queen Alexandra Hospital; Haematology and Oncology Centre, Portsmouth
  - Southampton General Hospital; Medical Oncology, Southampton
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton
  - Singleton Hospital; Pharmacy, Swansea
  - Great Western;Department of Haematology, Swindon
  - Royal Cornwall Hospital; Haematology Clinic, Truro

REFERENCES:
- [Derived] Pott C, Jurinovic V, Trotman J, Kehden B, Unterhalt M, Herold M, Jagt RV, Janssens A, Kneba M, Mayer J, Young M, Schmidt C, Knapp A, Nielsen T, Brown H, Spielewoy N, Harbron C, Bottos A, Mundt K, Marcus R, Hiddemann W, Hoster E. Minimal Residual Disease Status Predicts Outcome in Patients With Previously Untreated Follicular Lymphoma: A Prospective Analysis of the Phase III GALLIUM Study. J Clin Oncol. 2024 Feb 10;42(5):550-561. doi: 10.1200/JCO.23.00838. Epub 2023 Dec 14. PMID 38096461
- [Derived] Casulo C, Herold M, Hiddemann W, Iyengar S, Marcus RE, Seymour JF, Launonen A, Knapp A, Nielsen TG, Mir F. Risk Factors for and Outcomes of Follicular Lymphoma Histological Transformation at First Progression in the GALLIUM Study. Clin Lymphoma Myeloma Leuk. 2023 Jan;23(1):40-48. doi: 10.1016/j.clml.2022.09.003. Epub 2022 Oct 4. PMID 36379880
- [Derived] Hong X, Song Y, Shi Y, Zhang Q, Guo W, Wu G, Li J, Feng J, Kinkolykh A, Knapp A, Lin T. Efficacy and safety of obinutuzumab for the first-line treatment of follicular lymphoma: a subgroup analysis of Chinese patients enrolled in the phase III GALLIUM study. Chin Med J (Engl). 2021 Sep 16;135(4):433-440. doi: 10.1097/CM9.0000000000001737. PMID 35194005
- [Derived] Strefford JC, Nowicka M, Hargreaves CE, Burton C, Davies A, Ganderton R, Hiddemann W, Iriyama C, Klapper W, Latham KV, Martelli M, Mir F, Parker H, Potter KN, Rose-Zerilli MJJ, Sehn LH, Trneny M, Vitolo U, Bolen CR, Klein C, Knapp A, Oestergaard MZ, Cragg MS. Single-nucleotide Fcgamma receptor polymorphisms do not impact obinutuzumab/rituximab outcome in patients with lymphoma. Blood Adv. 2021 Aug 10;5(15):2935-2944. doi: 10.1182/bloodadvances.2020003985. PMID 34323957
- [Derived] Davies A, Trask P, Demeter J, Florschutz A, Hanel M, Kinoshita T, Pettengell R, Quach H, Robinson S, Sadullah S, Sancho JM, Udvardy M, Witzens-Harig M, Knapp A, Liu W. Health-related quality of life in the phase III GALLIUM study of obinutuzumab- or rituximab-based chemotherapy in patients with previously untreated advanced follicular lymphoma. Ann Hematol. 2020 Dec;99(12):2837-2846. doi: 10.1007/s00277-020-04021-6. Epub 2020 Apr 20. PMID 32314038
- [Derived] Klanova M, Oestergaard MZ, Trneny M, Hiddemann W, Marcus R, Sehn LH, Vitolo U, Bazeos A, Goede V, Zeuner H, Knapp A, Sahin D, Spielewoy N, Bolen CR, Cardona A, Klein C, Venstrom JM, Nielsen T, Fingerle-Rowson G. Prognostic Impact of Natural Killer Cell Count in Follicular Lymphoma and Diffuse Large B-cell Lymphoma Patients Treated with Immunochemotherapy. Clin Cancer Res. 2019 Aug 1;25(15):4634-4643. doi: 10.1158/1078-0432.CCR-18-3270. Epub 2019 May 3. PMID 31053601
- [Derived] Kusumoto S, Arcaini L, Hong X, Jin J, Kim WS, Kwong YL, Peters MG, Tanaka Y, Zelenetz AD, Kuriki H, Fingerle-Rowson G, Nielsen T, Ueda E, Piper-Lepoutre H, Sellam G, Tobinai K. Risk of HBV reactivation in patients with B-cell lymphomas receiving obinutuzumab or rituximab immunochemotherapy. Blood. 2019 Jan 10;133(2):137-146. doi: 10.1182/blood-2018-04-848044. Epub 2018 Oct 19. PMID 30341058
- [Derived] Trotman J, Barrington SF, Belada D, Meignan M, MacEwan R, Owen C, Ptacnik V, Rosta A, Fingerle-Rowson GR, Zhu J, Nielsen T, Sahin D, Hiddemann W, Marcus RE, Davies A; PET investigators from the GALLIUM study. Prognostic value of end-of-induction PET response after first-line immunochemotherapy for follicular lymphoma (GALLIUM): secondary analysis of a randomised, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1530-1542. doi: 10.1016/S1470-2045(18)30618-1. Epub 2018 Oct 8. PMID 30309758
- [Derived] Hiddemann W, Barbui AM, Canales MA, Cannell PK, Collins GP, Durig J, Forstpointner R, Herold M, Hertzberg M, Klanova M, Radford J, Seymour JF, Tobinai K, Trotman J, Burciu A, Fingerle-Rowson G, Wolbers M, Nielsen T, Marcus RE. Immunochemotherapy With Obinutuzumab or Rituximab for Previously Untreated Follicular Lymphoma in the GALLIUM Study: Influence of Chemotherapy on Efficacy and Safety. J Clin Oncol. 2018 Aug 10;36(23):2395-2404. doi: 10.1200/JCO.2017.76.8960. Epub 2018 Jun 1. PMID 29856692
- [Derived] Marcus R, Davies A, Ando K, Klapper W, Opat S, Owen C, Phillips E, Sangha R, Schlag R, Seymour JF, Townsend W, Trneny M, Wenger M, Fingerle-Rowson G, Rufibach K, Moore T, Herold M, Hiddemann W. Obinutuzumab for the First-Line Treatment of Follicular Lymphoma. N Engl J Med. 2017 Oct 5;377(14):1331-1344. doi: 10.1056/NEJMoa1614598. PMID 28976863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 177 centers in 18 countries.
Pre-assignment Details: Eleven participants withdrew from the study after randomization but prior to receiving study treatment.
Groups:
- Rituximab+Chemotherapy - Induction Period: Participants received either 8 cycles of rituximab along with 6 cycles of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) (21-day cycle) or 8 cycles of rituximab along with 8 cycles of cyclophosphamide, vincristine, and prednisone (CVP) (21-day cycles) or 6 cycles of rituximab along with 6 cycles of bendamustine (28-day cycle) during induction period. The chemotherapy regimen (CHOP or CVP or bendamustine) for individual participant was chosen by the site prior to initiation of the study.
- Obinutuzumab+Chemotherapy - Induction Period: Participants received either 8 cycles of obinutuzumab along with 6 cycles of CHOP (21-day cycle) or 8 cycles of obinutuzumab along with 8 cycles of CVP (21-day cycles) or 6 cycles of obinutuzumab along with 6 cycles of bendamustine (28-day cycle) during induction period. The chemotherapy regimen (CHOP or CVP or bendamustine) for individual participant was chosen by the site prior to initiation of the study.
- Rituximab+Chemotherapy - Maintenance Period: The induction period was followed by either a maintenance or observation period for responders or non-responders, respectively. Responders received rituximab monotherapy every 2 months for 2 years during the maintenance period.
- Obinutuzumab+Chemotherapy - Maintenance Period: The induction period was followed by either a maintenance or observation period for responders or non-responders, respectively. Responders received obinutuzumab monotherapy every 2 months for 2 years during the maintenance period.
- Rituximab+Chemotherapy - Observation Period: Rituximab+Chemotherapy - Observation: The induction period was followed by either a maintenance or observation period for responders or non-responders, respectively. Non-responders received no protocol specified treatment during the 2-year observation period.
- Obinutuzumab+Chemotherapy - Observation Period: Obinutuzumab+Chemotherapy - Observation: The induction period was followed by either a maintenance or observation period for responders or non-responders, respectively. Non-responders received no protocol specified treatment during the 2-year observation period.
- Rituximab+Chemotherapy - Follow-Up Period; Obinutuzumab+Chemotherapy - Follow-Up Period: Finally, participants were followed during a 5-year follow-up period.
Period: Induction Period
Arm/Group | Rituximab+Chemotherapy - Induction Period | Obinutuzumab+Chemotherapy - Induction Period | Rituximab+Chemotherapy - Maintenance Period | Obinutuzumab+Chemotherapy - Maintenance Period | Rituximab+Chemotherapy - Observation Period | Obinutuzumab+Chemotherapy - Observation Period | Rituximab+Chemotherapy - Follow-Up Period | Obinutuzumab+Chemotherapy - Follow-Up Period
Started | 699 | 702 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 641 | 646 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 58 | 56 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 23 | 26 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 15 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomised but not treated | 4 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance/Observation Period
Arm/Group | Rituximab+Chemotherapy - Induction Period | Obinutuzumab+Chemotherapy - Induction Period | Rituximab+Chemotherapy - Maintenance Period | Obinutuzumab+Chemotherapy - Maintenance Period | Rituximab+Chemotherapy - Observation Period | Obinutuzumab+Chemotherapy - Observation Period | Rituximab+Chemotherapy - Follow-Up Period | Obinutuzumab+Chemotherapy - Follow-Up Period
Started | 0 | 0 | 612 | 624 | 12 | 11 | 0 | 0
Completed | 0 | 0 | 451 | 475 | 12 | 10 | 0 | 0
Not Completed | 0 | 0 | 161 | 149 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 53 | 66 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 4 | 3 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 4 | 7 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 14 | 19 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 72 | 40 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 5 | 0 | 0 | 0 | 0
Period: Follow-Up Period
Arm/Group | Rituximab+Chemotherapy - Induction Period | Obinutuzumab+Chemotherapy - Induction Period | Rituximab+Chemotherapy - Maintenance Period | Obinutuzumab+Chemotherapy - Maintenance Period | Rituximab+Chemotherapy - Observation Period | Obinutuzumab+Chemotherapy - Observation Period | Rituximab+Chemotherapy - Follow-Up Period | Obinutuzumab+Chemotherapy - Follow-Up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 554 | 602
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 324 | 367
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 230 | 235
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 30
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 15
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 9
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 21
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 15
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 126 | 106
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 32
Not completed — No reason provided | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to treat (ITT) population was defined as all randomized participants grouped according to their randomized treatment arm regardless of what treatments were actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab+Chemotherapy - Induction Period | Obinutuzumab+Chemotherapy - Induction Period | Total
Number analyzed (Participants) | 699 | 702 | 1401
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.3) | 58.9 (11.6) | 58.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374 | 365 | 739
  Male | 325 | 337 | 662
Age Continuous in Follicular Lymphoma Sub-Population [Mean (Standard Deviation); unit: years] — Age continuous for participants with follicular lymphoma (FL) in each arm, who encompassed the population for the primary outcome measure. The FL ITT included participants in the ITT population with follicular histology (n=601 in each arm).
  years | 57.7 (12.2) | 58.2 (11.5) | 57.9 (11.9)
Gender in Follicular Lymphoma Sub-Population [Count of Participants; unit: Participants] — Gender of participants with follicular lymphoma, who encompassed the population for the primary outcome measure. The FL ITT included participants in the ITT population with follicular histology (n=601 for each arm). Population: As this is a sub-population, the numbers analyzed differ from the overall population numbers as not all are included here.
  Participants
    number analyzed (Participants) | 601 | 601 | 1202
    Female | 321 | 318 | 639
    Male | 280 | 283 | 563

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival in the Follicular Lymphoma Population, Investigator-Assessed
Description: Progression-free survival in participants with follicular lymphoma was defined as the time from randomization until the first documented day of disease progression or death from any cause, whichever occurred first, on the basis of investigator assessments according to the Revised Response Criteria for Malignant Lymphoma. Progression was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Tumor measurements were obtained by computed tomography (CT) or magnetic resonance imaging (MRI).
Time Frame: Baseline up to data cut-off (up to approximately 4 years and 7 months)
Population: The intent-to-treat follicular lymphoma population (FL ITT), defined as all randomized participants with follicular histology, where participants were grouped according to their randomized treatment arm regardless of what treatments were actually received.
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event | 24.0 | 16.8
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority or Other; p = 0.0012, Log Rank; Stratified by chemotherapy regimen and Follicular Lymphoma International Prognostic Index (FLIPI) risk group; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.51 to 0.85]

2. Secondary Outcome: Progression-Free Survival in the Follicular Lymphoma Population, Investigator-Assessed
Description: as for outcome 1
Time Frame: Baseline up to final analysis (up to 10 years)
Population: The FL ITT population was defined as all randomized participants with follicular histology, where participants were grouped according to their randomized treatment arm regardless of what treatments were actually received.
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event | 40.6 | 34.3
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority or Other; p = 0.0055, Log Rank; Stratified by chemotherapy regimen and Follicular Lymphoma International Prognostic Index (FLIPI) risk group; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.64 to 0.93]

3. Secondary Outcome: Progression-Free Survival in the Overall Study Population, Investigator-Assessed
Description: Progression-free survival in the overall study population was defined as the time from randomization until the first documented day of disease progression or death from any cause, whichever occurred first, on the basis of investigator assessments according to the Revised Response Criteria for Malignant Lymphoma. Progression was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Tumor measurements were obtained by CT/MRI.
Time Frame: Baseline up to data cut-off (up to approximately 5 years and 2 months)
Population: The ITT population defined as all randomized participants grouped according to their randomized treatment arm regardless of what treatments were actually received.
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 699 | 702
percentage of participants with event | 41.5 | 34.8
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.0028, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.65 to 0.91]

4. Secondary Outcome: Progression-Free Survival (Follicular Lymphoma Population), IRC-Assessed
Description: Progression-free survival in the participants with follicular lymphoma was defined as the time from randomization until the first documented day of disease progression or death from any cause, whichever occurred first, on the basis of IRC assessments according to the Revised Response Criteria for Malignant Lymphoma. Progression was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Tumor measurements were obtained by CT/MRI. In the first 170 patients with follicular lymphoma, an FDG-PET was mandatory where a PET scanner was available.
Time Frame: Baseline up to data cut-off (up to approximately 5 years and 2 months)
Population: The FL ITT population, defined as all randomized participants with follicular histology, where participants were grouped according to their randomized treatment arm regardless of what treatments were actually received.
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event | 23.5 | 18.0
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.0118, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.56 to 0.93]

5. Secondary Outcome: Progression-Free Survival (Overall Study Population), Assessed by Independent Review Committee (IRC)
Description: Progression-free survival in the overall study population was defined as the time from randomization until the first documented day of disease progression or death from any cause, whichever occurred first, on the basis of IRC assessments according to the Revised Response Criteria for Malignant Lymphoma. Progression was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Tumor measurements were obtained by CT/MRI.
Time Frame: Baseline up to data cut-off (up to approximately 5 years and 2 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 699 | 702
percentage of participants with event | 24.6 | 18.4
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.0038, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI [0.57 to 0.90]

6. Secondary Outcome: Overall Response (Follicular Lymphoma Population), Investigator-Assessed
Description: Overall response in the follicular lymphoma population was defined as percentage of participants with PR or complete response CR determined on the basis of investigator assessments with the use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI with and without PET. CR was defined as disappearance of all target lesions; PR was defined as >=50% decrease target lesions in up to six dominant lesions identified at baseline, no new lesions and no increase in the size of the liver, spleen, or other nodes. Splenic and hepatic nodules must have regressed by >/= 50%. Overall Response (OR) = CR + PR.
Time Frame: Baseline up to end of induction period (up to approximately 7 months)
Population: as for outcome 4
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event
  Without PET: number analyzed (Participants) | 519 | 530
  Without PET | 86.4 | 88.2
  With PET: number analyzed (Participants) | 242 | 254
  With PET | 81.2 | 85.5
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Without PET; Test type: Superiority; p = 0.30, Log Rank; Absolute difference in % = 1.8, 95% CI 2-sided [-2.02 to 5.68]
Statistical Analysis 2: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; With PET; Test type: Superiority; p = 0.17, Log Rank; Absolute difference in % = 4.3, 95% CI 2-sided [-1.8 to 10.5]

7. Secondary Outcome: Overall Response (Overall Study Population), Investigator-Assessed
Description: Overall response in the overall study population was defined as percentage of participants with partial response (PR) or complete response (CR) determined on the basis of investigator assessments with the use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI with or without positron emission tomography (PET). CR was defined as disappearance of all target lesions; PR was defined as >=50% decrease target lesions in up to six dominant lesions identified at baseline, no new lesions and no increase in the size of the liver, spleen, or other nodes. Splenic and hepatic nodules must have regressed by >/= 50%; Overall Response (OR) = CR + PR.
Time Frame: Baseline up to end of induction period (up to approximately 7 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 699 | 702
percentage of participants with event
  Without PET: number analyzed (Participants) | 599 | 613
  Without PET | 85.7 | 87.3
  With PET: number analyzed (Participants) | 270 | 274
  With PET | 81.8 | 85.4
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Without PET; Test type: Superiority; p = 0.33, Log Rank; Absolute difference in % = 1.6, 95% CI 2-sided [-2.0 to 5.3]
Statistical Analysis 2: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; With PET; Test type: Superiority; p = 0.17, Log Rank; Absolute difference in % = 3.5, 95% CI 2-sided [-2.3 to 9.4]

8. Secondary Outcome: Complete Response (Follicular Lymphoma Population), Investigator-Assessed
Description: Percentage of participants with complete response in the follicular lymphoma population was determined on the basis of investigator assessments with the use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI with or without PET. CR was defined as disappearance of all target lesions.
Time Frame: Baseline up to end of induction period (up to approximately 7 months)
Population: as for outcome 4
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event
  Without PET: number analyzed (Participants) | 145 | 112
  Without PET | 24.1 | 18.6
  With PET: number analyzed (Participants) | 169 | 184
  With PET | 56.7 | 62.0
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Without PET; Test type: Superiority; p = 0.02, Log Rank; Absolute difference in % = -5.5, 95% CI 2-sided [-10.2 to -0.78]
Statistical Analysis 2: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; With PET; Test type: Superiority; p = 0.32, Log Rank; Absolute difference in % = 5.2, 95% CI 2-sided [-2.8 to 13.3]

9. Secondary Outcome: Complete Response (Overall Study Population), Investigator-Assessed
Description: Percentage of participants with complete response in the overall study population was determined on the basis of investigator assessments with the use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI with or without PET. CR was defined as disappearance of all target lesions.
Time Frame: Baseline up to end of induction period (up to approximately 7 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 699 | 702
percentage of participants with event
  Without PET: number analyzed (Participants) | 163 | 129
  Without PET | 23.3 | 18.4
  With PET: number analyzed (Participants) | 188 | 196
  With PET | 57.0 | 61.1
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Without PET; Test type: Superiority; p = 0.02, Log Rank; Absolute difference in % = -4.9, 95% CI [-9.3 to 0.6]
Statistical Analysis 2: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; With PET; Test type: Superiority; p = 0.33, Log Rank; Absolute difference in % = 4.1, 95% CI [-3.6 to 11.8]

10. Secondary Outcome: Overall Response (Follicular Lymphoma Population), IRC-Assessed
Description: Overall response in the follicular lymphoma population was defined as percentage of participants with PR or complete response CR determined on the basis of IRC assessments with the use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI with or without PET. CR was defined as disappearance of all target lesions; PR was defined as >=50% decrease target lesions in up to six dominant lesions identified at baseline, no new lesions and no increase in the size of the liver, spleen, or other nodes. Splenic and hepatic nodules must have regressed by >/= 50%. Overall Response (OR) = CR + PR.
Time Frame: Baseline up to end of induction period (up to approximately 7 months)
Population: as for outcome 4
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event
  Without PET: number analyzed (Participants) | 529 | 549
  Without PET | 88.0 | 91.3
  With PET: number analyzed (Participants) | 254 | 263
  With PET | 85.2 | 88.6
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Without PET; Test type: Superiority; p = 0.052, Log Rank; Absolute difference in % = 3.3, 95% CI 2-sided [-0.19 to 6.85]
Statistical Analysis 2: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; With PET; Test type: Superiority; p = 0.30, Log Rank; Absolute difference in % = 3.3, 95% CI 2-sided [-2.3 to 8.9]

11. Secondary Outcome: Overall Response (Overall Study Population), IRC-Assessed
Description: Overall response in the overall study population was defined as percentage of participants with PR or CR determined on the basis of IRC assessments with the use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI with or without PET. CR was defined as disappearance of all target lesions; PR was defined as >=50% decrease target lesions in up to six dominant lesions identified at baseline, no new lesions and no increase in the size of the liver, spleen, or other nodes. Splenic and hepatic nodules must have regressed by >/= 50%; Overall Response (OR) = CR + PR.
Time Frame: Baseline up to end of induction period (up to approximately 7 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 699 | 702
percentage of participants with event
  Without PET: number analyzed (Participants) | 606 | 631
  Without PET | 86.7 | 89.9
  With PET: number analyzed (Participants) | 330 | 321
  With PET | 83.3 | 87.2
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Without PET; Test type: Superiority; p = 0.049, Log Rank; Absolute difference in % = 3.2, 95% CI 2-sided [-0.3 to 6.6]
Statistical Analysis 2: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; With PET; Test type: Superiority; p = 0.22, Log Rank; Absolute difference in % = 3.9, 95% CI 2-sided [-1.7 to 9.5]

12. Secondary Outcome: Complete Response (Follicular Lymphoma Population), IRC-Assessed
Description: Percentage of participants with complete response in the follicular lymphoma population was determined on the basis of IRC assessments with the use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI with or without PET. CR was defined as disappearance of all target lesions.
Time Frame: Baseline up to end of induction period (up to approximately 7 months)
Population: as for outcome 4
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event
  Without PET: number analyzed (Participants) | 161 | 171
  Without PET | 26.8 | 28.5
  With PET: number analyzed (Participants) | 178 | 212
  With PET | 59.7 | 71.4
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Without PET; Test type: Superiority; p = 0.58, Log Rank; Absolute difference in % = 1.7, 95% CI 2-sided [-3.5 to 6.8]
Statistical Analysis 2: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.006, Log Rank; Absolute difference in % = 11.7, 95% CI 2-sided [3.9 to 19.4]

13. Secondary Outcome: Complete Response (Overall Study Population), IRC-Assessed
Description: Percentage of participants with complete response in the overall study population was determined on the basis of IRC assessments with the use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI with or without PET. CR was defined as disappearance of all target lesions.
Time Frame: Baseline up to end of induction period (up to approximately 7 months)]
Population: as for outcome 3
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 699 | 702
percentage of participants with event
  Without PET: number analyzed (Participants) | 184 | 190
  Without PET | 26.3 | 27.1
  With PET: number analyzed (Participants) | 196 | 223
  With PET | 59.4 | 69.5
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Without PET; Test type: Superiority; p = 0.80, Log Rank; Absolute difference in % = 0.7, 95% CI 2-sided [-4.0 to 5.5]
Statistical Analysis 2: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; With PET; Test type: Superiority; p = 0.009, Log Rank; Absolute difference in % = 10.1, 95% CI [2.6 to 17.6]

14. Secondary Outcome: Overall Survival (Follicular Lymphoma Population)
Description: Overall survival in the follicular lymphoma population was defined as the time from the date of randomization to the date of death from any cause. Reported is the percentage of participants with event.
Time Frame: Baseline up to 10 years
Population: as for outcome 4
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event | 14.3 | 12.6
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.3577, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI [0.63 to 1.18]

15. Secondary Outcome: Overall Survival (Overall Study Population)
Description: Overall survival in the overall study population was defined as the time from the date of randomization to the date of death from any cause. Reported is the percentage of participants with event.
Time Frame: Baseline up to data cut-off (up to approximately 5 years and 2 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 699 | 702
percentage of participants with event | 10.2 | 8.4
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.25, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI [0.58 to 1.16]

16. Secondary Outcome: Event-Free Survival (Follicular Lymphoma Population)
Description: Event-free survival in the follicular lymphoma population was defined as the time from the date of randomization to the date to disease progression/relapse, death from any cause, or initiation of a new anti-lymphoma treatment (NALT) on the basis of investigator assessment assessments with the use of Revised Response Criteria for Malignant Lymphoma. Disease progression/relapse was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Tumor measurements were obtained by CT/MRI. Reported is the percentage of participants with an event.
Time Frame: Baseline up to 10 years
Population: as for outcome 4
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event | 42.9 | 35.8
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.0015, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.62 to 0.89]

17. Secondary Outcome: Event-Free Survival (Overall Study Population)
Description: Event-free survival in the overall study population was defined as the time from the date of randomization to the date to disease progression/relapse, death from any cause, or initiation of a new anti-lymphoma treatment (NALT) on the basis of investigator assessment assessments with the use of Revised Response Criteria for Malignant Lymphoma. Disease progression/relapse was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Tumor measurements were obtained by CT/MRI. Reported is the percentage of participants with event.
Time Frame: Baseline up to data cut-off (up to approximately 5 years and 2 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 699 | 702
percentage of participants with event | 30.6 | 22.6
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI [0.56 to 0.85]

18. Secondary Outcome: Disease-Free Survival (Follicular Lymphoma Population)
Description: Disease-free survival in the follicular lymphoma population was defined as the time from the date of the first occurrence of a documented CR to the date of disease progression/ relapse, or death from any cause for the subgroup of participants with a response of CR at any time prior to NALT on the basis of investigator assessments with the use of Revised Response Criteria for Malignant Lymphoma (RRCML). Tumor assessments were performed with CT/MRI. CR was defined as disappearance of all target lesions. Progression/relapse was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Reported is the percentage of participants with event.
Time Frame: From first occurrence of documented CR to data cut-off (up to approximately 5 years and 2 months)
Population: Participants with CR within the FL ITT population were included in the analysis.The FL ITT population, defined as all randomized participants with follicular histology, where participants were grouped according to their randomized treatment arm regardless of what treatments were actually received.
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 330 | 355
percentage of participants with event | 27.9 | 26.3
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.71 to 1.27]

19. Secondary Outcome: Disease-Free Survival (Overall Study Population)
Description: Disease-free survival in the overall study population was defined as the time from the date of the first occurrence of a documented CR to the date of disease progression/ relapse, or death from any cause for the subgroup of participants with a response of CR at any time prior to NALT on the basis of investigator assessments with the use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI. CR was defined as disappearance of all target lesions. Progression/relapse was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Reported is the percentage of participants with event.
Time Frame: From first occurrence of documented CR to data cut-off (up to approximately 5 years and 2 months)
Population: Participants with CR within the ITT population were included in the analysis.The ITT population was defined as all randomized participants grouped according to their randomized treatment arm regardless of what treatments were actually received.
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 320 | 343
percentage of participants with event | 14.9 | 11.2
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.50 to 1.19]

20. Secondary Outcome: Duration of Response (DOR) (Follicular Lymphoma Population), Investigator-Assessed
Description: DOR was defined as the time from first occurrence of a documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR any time prior to NALT based on RRCML. Tumor assessments were performed with CT/MRI. CR was defined as disappearance of all target lesions. PR was defined as >/=50% decrease target lesions in up to six dominant lesions identified at baseline, no new lesions and no increase in the size of the liver, spleen, or other nodes. Splenic and hepatic nodules must have regressed by >/= 50%. Progression/relapse was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm.
Time Frame: From first occurrence of documented CR or PR to data cut-off (up to approximately 5 years and 2 months)
Population: Participants with CR or PR within the FL ITT population were included in the analysis.The FL ITT population, defined as all randomized participants with follicular histology, where participants were grouped according to their randomized treatment arm regardless of what treatments were actually received.
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 568 | 571
percentage of participants with event | 39.3 | 33.3
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.63 to 0.93]

21. Secondary Outcome: Duration of Response (DOR) (Overall Study Population), Investigator-Assessed
Description: as for outcome 20
Time Frame: From first occurrence of documented CR or PR to data cut-off (up to approximately 4 years and 7 months)
Population: Participants with CR or PR within the ITT population were included in the analysis. The ITT population defined as all randomized participants grouped according to their randomized treatment arm regardless of what treatments were actually received.
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 656 | 659
percentage of participants with event | 25.5 | 18.7
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.69, 95% CI [0.55 to 0.88]

22. Secondary Outcome: Time to Next Anti-Lymphoma Treatment (Follicular Lymphoma Population)
Description: Time to next anti-lymphoma treatment was defined as the time from the date of randomization to the start date of the next anti-lymphoma treatment or death from any cause. Reported is the percentage of participants with event.
Time Frame: Baseline up to 10 years
Population: as for outcome 4
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 601 | 601
percentage of participants with event | 34.8 | 26.6
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.001, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.58 to 0.87]

23. Secondary Outcome: Time to Next Anti-Lymphoma Treatment (Overall Study Population)
Description: as for outcome 22
Time Frame: Baseline up to data cut-off (up to approximately 5 years and 2 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants with event
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 699 | 702
percentage of participants with event | 21.6 | 15.7
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority; p = 0.004, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI [0.54 to 0.89]

24. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to 10 years
Population: The safety analysis population included all participants who received any amount of any study drug and participants were analyzed according to the treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 692 | 698
percentage of participants | 99.6 | 99.9

25. Secondary Outcome: Change From Baseline in All Domains of FACT-G (Follicular Lymphoma Population)
Description: FACT-G consists of the following 4 FACT-Lym sub-questionnaires: Physical Well-being (range: 0-28), Social/Family Well-being (range: 0-28), Emotional Well-being (range: 0-24) and Functional Well-being (range: 0-28). Higher scores indicate better outcomes. A positive change from baseline indicates improvement. Maint = Maintenance period.
Time Frame: Baseline (Induction Cycle 1, Day 1), data cut-off (up to approximately 5 years and 2 months)
Population: The FL ITT population was defined as all randomized participants with follicular histology grouped according to their randomized treatment arm regardless of what treatments were actually received.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Rituximab+Chemotherapy: Participants received either 8 cycles of rituximab along with 6 cycles of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) (21-day cycle) or 8 cycles of rituximab along with 8 cycles of cyclophosphamide, vincristine, and prednisone (CVP) (21-day cycles) or 6 cycles of rituximab along with 6 cycles of bendamustine (28-day cycle) during the induction period. The induction period was followed by either a maintenance or observation period for responders or non-responders, respectively. Responders received rituximab monotherapy every 2 months for 2 years during the maintenance period. Non-responders received no protocol specified treatment during the 2-year observation period. Finally, participants were followed during a 5-year follow-up period. The chemotherapy regimen (CHOP or CVP or bendamustine) for individual participant was chosen by the site prior to initiation of the study.
- Obinutuzumab+Chemotherapy: Participants received either 8 cycles of obinutuzumab along with 6 cycles of CHOP (21-day cycle) or 8 cycles of obinutuzumab along with 8 cycles of CVP (21-day cycles) or 6 cycles of obinutuzumab along with 6 cycles of bendamustine (28-day cycle) during induction period. The induction period was followed by either a maintenance or observation period for responders or non-responders, respectively. Responders received obinutuzumab monotherapy every 2 months for 2 years during the maintenance period. Non-responders received no protocol specified treatment during the 2-year observation period. Finally, participants were followed during a 5-year follow-up period. The chemotherapy regimen (CHOP or CVP or bendamustine) for individual participant was chosen by the site prior to initiation of the study.
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 557 | 566
units on a scale
  Physical Well-being (PW), Baseline | 23.36 (4.77) | 23.14 (4.85)
  PW Change, Cycle 3, Day 1: number analyzed (Participants) | 511 | 496
  PW Change, Cycle 3, Day 1 | -0.91 (4.54) | -0.21 (4.59)
  PW Change, End Induction: number analyzed (Participants) | 482 | 480
  PW Change, End Induction | -0.06 (4.83) | 0.56 (5.14)
  PW Change, Maint Month 2: number analyzed (Participants) | 362 | 398
  PW Change, Maint Month 2 | 0.83 (4.76) | 1.42 (5.09)
  PW Change, Maint Month 12: number analyzed (Participants) | 362 | 406
  PW Change, Maint Month 12 | 1.14 (4.29) | 1.34 (4.74)
  PW Change, End Maint: number analyzed (Participants) | 411 | 437
  PW Change, End Maint | 0.88 (4.54) | 1.33 (5.00)
  Social/Family Well-being , Baseline: number analyzed (Participants) | 555 | 563
  Social/Family Well-being , Baseline | 22.84 (4.92) | 23.28 (4.77)
  S/FW Change, Cycle 3 Day 1: number analyzed (Participants) | 506 | 492
  S/FW Change, Cycle 3 Day 1 | -0.52 (4.03) | -0.67 (3.92)
  S/FW Change, End Induction: number analyzed (Participants) | 482 | 475
  S/FW Change, End Induction | -0.46 (4.77) | -0.56 (5.00)
  S/FW Change, Maint Month 2: number analyzed (Participants) | 359 | 396
  S/FW Change, Maint Month 2 | -0.39 (4.72) | -0.67 (4.68)
  S/FW Change, Maint Month 12: number analyzed (Participants) | 359 | 403
  S/FW Change, Maint Month 12 | -0.61 (5.56) | -0.97 (5.34)
  S/FW Change, End Maint: number analyzed (Participants) | 410 | 436
  S/FW Change, End Maint | -0.93 (5.67) | -0.71 (5.54)
  Emotional Well-being (EW), Baseline: number analyzed (Participants) | 556 | 563
  Emotional Well-being (EW), Baseline | 17.64 (4.19) | 17.87 (4.13)
  EW Change, Cycle 3 Day 1: number analyzed (Participants) | 503 | 490
  EW Change, Cycle 3 Day 1 | 1.49 (3.40) | 1.35 (3.35)
  EW Change, End Induction: number analyzed (Participants) | 478 | 476
  EW Change, End Induction | 1.16 (3.90) | 1.14 (3.87)
  EW Change, Maint Month 2: number analyzed (Participants) | 359 | 396
  EW Change, Maint Month 2 | 1.77 (3.88) | 1.49 (4.16)
  EW Change, Maint Month 12: number analyzed (Participants) | 360 | 402
  EW Change, Maint Month 12 | 1.45 (3.92) | 1.46 (3.88)
  EW Change, End Maint: number analyzed (Participants) | 405 | 435
  EW Change, End Maint | 1.43 (3.98) | 1.49 (3.99)
  Functional Well-being (FW), Baseline: number analyzed (Participants) | 556 | 563
  Functional Well-being (FW), Baseline | 18.66 (6.19) | 18.76 (5.98)
  FW Change, Cycle 3 Day 1: number analyzed (Participants) | 504 | 488
  FW Change, Cycle 3 Day 1 | -0.30 (5.30) | -0.07 (5.24)
  FW Change, End Induction: number analyzed (Participants) | 480 | 476
  FW Change, End Induction | 0.44 (5.63) | 0.93 (5.85)
  FW Change, Maint Month 2: number analyzed (Participants) | 359 | 396
  FW Change, Maint Month 2 | 1.04 (5.31) | 1.25 (6.02)
  FW Change, Maint Month 12: number analyzed (Participants) | 360 | 402
  FW Change, Maint Month 12 | 1.84 (5.54) | 1.65 (5.95)
  FW Change, End Maint: number analyzed (Participants) | 406 | 436
  FW Change, End Maint | 1.40 (6.12) | 1.72 (6.16)

26. Secondary Outcome: Change From Baseline in FACT-Lym Total Outcome Index (TOI) Score (Follicular Lymphoma Population)
Description: The FACT-Lym TOI Score for the follicular lymphoma population was derived from the following 3 individual FACT-Lym questionnaire subscale scores: Physical Well-being (range: 0-28), Functional Well-being (range: 0-28) and Lymphoma (range: 0-60). The FACT-Lym TOI Score is the sum of the 3 individual subscales (range 0-116). Higher scores indicate better outcomes. A positive change from baseline indicates an improvement.
Time Frame: Baseline (Induction Cycle 1, Day 1), data cut-off (up to approximately 5 years and 2 months)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 559 | 567
units on a scale
  TOI Score, Baseline | 86.61 (18.16) | 86.94 (18.05)
  TOI Score Change, Cycle 3 Day 1: number analyzed (Participants) | 514 | 497
  TOI Score Change, Cycle 3 Day 1 | 0.46 (15.03) | 2.18 (15.95)
  TOI Score Change, End Induction: number analyzed (Participants) | 485 | 481
  TOI Score Change, End Induction | 2.91 (17.00) | 4.57 (16.71)
  TOI Score Change, Maint M2: number analyzed (Participants) | 363 | 400
  TOI Score Change, Maint M2 | 6.22 (16.16) | 7.17 (16.57)
  TOI Score Change, Maint M12: number analyzed (Participants) | 362 | 408
  TOI Score Change, Maint M12 | 7.61 (15.62) | 7.20 (16.75)
  TOI Score Change, End Maint: number analyzed (Participants) | 412 | 440
  TOI Score Change, End Maint | 6.23 (17.06) | 7.44 (16.96)

27. Secondary Outcome: Change From Baseline in FACT-Lym Individual Subscale Lymphoma Score (Follicular Population)
Description: The FACT-Lym Individual Subscale Lymphoma Score for the follicular lymphoma population was derived from the Lymphoma subscale questionnaire (range: 0-60). Higher scores indicate better outcomes. A positive change from baseline indicates an improvement.
Time Frame: Baseline (Induction Cycle 1, Day 1), data cut-off (up to approximately 5 years and 2 months)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 556 | 563
units on a scale
  Lymphoma, Baseline | 45.01 (9.37) | 45.54 (9.29)
  Lymphoma Change, Cycle 3 Day 1: number analyzed (Participants) | 509 | 491
  Lymphoma Change, Cycle 3 Day 1 | 2.04 (7.18) | 2.71 (7.46)
  Lymphoma Change, End Induction: number analyzed (Participants) | 477 | 478
  Lymphoma Change, End Induction | 2.99 (8.63) | 3.01 (8.36)
  Lymphoma Change, Maint Month 2: number analyzed (Participants) | 360 | 395
  Lymphoma Change, Maint Month 2 | 4.80 (8.29) | 4.52 (8.32)
  Lymphoma Change, Maint Month 12: number analyzed (Participants) | 360 | 404
  Lymphoma Change, Maint Month 12 | 4.93 (8.34) | 4.27 (8.31)
  Lymphoma Change, End Maint: number analyzed (Participants) | 407 | 438
  Lymphoma Change, End Maint | 4.31 (8.81) | 4.57 (8.54)

28. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) Total Score (Follicular Population)
Description: The FACT-Lym Total Score for the follicular lymphoma population was derived from the following 5 individual FACT-Lym questionnaire subscale scores: Physical Well-being (range: 0-28), Social/Family Well-being (range: 0-28), Emotional Well-being (range: 0-24),Functional Well-being (range: 0-28) and Lymphoma (range: 0-60). The FACT-Lym Total Score is the sum of all 5 individual subscales (range 0-168). Higher scores indicate better outcomes. A positive change from baseline indicates an improvement.
Time Frame: Baseline (Induction Cycle 1, Day 1), data cut-off (up to approximately 5 years and 2 months)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 552 | 559
units on a scale
  Total Score, Baseline | 127.40 (22.43) | 128.42 (22.16)
  Total Score Change, Cycle 3 Day 1: number analyzed (Participants) | 499 | 484
  Total Score Change, Cycle 3 Day 1 | 1.98 (17.01) | 3.21 (17.12)
  Total Score Change, End Induction: number analyzed (Participants) | 471 | 471
  Total Score Change, End Induction | 4.18 (19.75) | 5.10 (20.03)
  Total Score Change, Maint Month 2: number analyzed (Participants) | 356 | 392
  Total Score Change, Maint Month 2 | 8.40 (19.16) | 8.13 (19.80)
  Total Score Change, Maint Month 12: number analyzed (Participants) | 358 | 396
  Total Score Change, Maint Month 12 | 8.87 (19.31) | 7.90 (19.55)
  Total Score Change, End Maint: number analyzed (Participants) | 401 | 433
  Total Score Change, End Maint | 7.43 (19.88) | 8.80 (20.57)

29. Secondary Outcome: Change From Baseline in Euro-Quality of Life-5 Dimensions (EQ-5D) Questionnaire Summary Score (Follicular Lymphoma Population) During Induction Phase
Description: The EQ-5D is a quality of life questionnaire with five questions, each with three categories (no problem, moderate problem, severe problems) and a visual analogue scale (VAS) from 0 (worst possible health state) to 100 (best possible health state. Summary score ranges from 0 to 1. Higher scores indicate better outcomes. A positive change from baseline indicates an improvement. Completion (Compl) includes completion visit and early termination visit. Maintenance/Observation is indicated as Maint/Obs.
Time Frame: Induction: Cycle 1 Day 1 (Baseline), Cycle 3 Day 1, End of Induction (up to 7 months); Maintenance: 2, 12 months after Day 1 of last induction cycle, Follow-up: every year up to data cut-off (up to 5 years and 2 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 558 | 559
units on a scale
  Baseline Induction | 0.80 (0.24) | 0.81 (0.21)
  Change Baseline, Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Change Baseline, Cycle 3 Day 1: number analyzed (Participants) | 505 | 487
  Change Baseline, Cycle 3 Day 1 | 0.03 (0.21) | 0.03 (0.20)
  Change Baseline, Induction Compl: number analyzed (Participants) | 468 | 466
  Change Baseline, Induction Compl | 0.04 (0.23) | 0.03 (0.22)
  Change Baseline, Maint/Obs Month 2: number analyzed (Participants) | 348 | 377
  Change Baseline, Maint/Obs Month 2 | 0.05 (0.23) | 0.06 (0.22)
  Change from Baseline, Maint/Obs Month 12: number analyzed (Participants) | 2 | 1
  Change from Baseline, Maint/Obs Month 12 | 0.00 (0.00) | -0.20 (NA) — NA = NE = Not estimable based on 1 participant evaluated
  Change Baseline, Maint/Obs Completion: number analyzed (Participants) | 0 | 1
  Change Baseline, Maint/Obs Completion |  | -0.10 (NA) — NA = NE = Not estimable based on 1 participant evaluated

30. Secondary Outcome: Change From Baseline in Euro-Quality of Life-5 Dimensions (EQ-5D) Questionnaire Summary Score (Follicular Lymphoma Population) During Maintenance/Observation Phase
Description: The EQ-5D is a quality of life questionnaire with five questions, each with three categories (no problem, moderate problem, severe problems) and a visual analogue scale (VAS) from 0 (worst possible health state) to 100 (best possible health state. Summary score ranges from 0 to 1 Higher scores indicate better outcomes. A positive change from baseline indicates an improvement. Maintenance/Observation is indicated as Maint/Obs. Completion includes completion visit and early termination visit.
Time Frame: as for outcome 29
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 536 | 547
units on a scale
  Change Baseline, Maint/Obs Month 2: number analyzed (Participants) | 11 | 14
  Change Baseline, Maint/Obs Month 2 | 0.04 (0.34) | 0.04 (0.14)
  Change Baseline, Maint/Obs Month 12 | 0.06 (0.24) | 0.06 (0.21)
  Change Baseline, Maint/Obs Completion: number analyzed (Participants) | 402 | 421
  Change Baseline, Maint/Obs Completion | 0.03 (0.23) | 0.05 (0.23)

31. Secondary Outcome: Change From Baseline in Euro-Quality of Life-5 Dimensions (EQ-5D) Questionnaire Summary Score (Follicular Lymphoma Population) During Follow Up Phase
Description: The EQ-5D is a quality of life questionnaire with five questions, each with three categories (no problem, moderate problem, severe problems) and a visual analogue scale (VAS) from 0 (worst possible health state) to 100 (best possible health state. Summary score ranges from 0 to 1. Higher scores indicate better outcomes. A positive change from baseline indicates an improvement. Maintenance/Observation is indicated as Maint/Obs in data categories. Completion includes completion visit and early termination visit.
Time Frame: Induction: Cycle 1 Day 1 (Baseline), Cycle 3 Day 1, End of Induction (up to 7 months); Maintenance: 2, 12 after Day 1 of last induction cycle, Follow-up: every year for up to data cut-off (up to 5 years and 2 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 563 | 564
units on a scale
  Change Baseline, Follow-Up Month 36: number analyzed (Participants) | 238 | 248
  Change Baseline, Follow-Up Month 36 | 0.05 (0.24) | 0.06 (0.23)
  Change Baseline, Follow-Up Month 48: number analyzed (Participants) | 73 | 80
  Change Baseline, Follow-Up Month 48 | 0.05 (0.20) | 0.06 (0.23)

ADVERSE EVENTS:
Time Frame: Baseline up to 10 years
Description: The safety analysis population included all participants who received any amount of any study drug and participants were analyzed according to the treatment received.
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
All-Cause Mortality (participants affected / at risk) | 111/692 | 104/698
Serious Adverse Events (participants affected / at risk) | 309/692 | 361/698
Other Adverse Events (participants affected / at risk) | 675/692 | 690/698
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab+Chemotherapy (N=692) | Obinutuzumab+Chemotherapy (N=698)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 6 (7)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 23 (31) | 36 (48)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HAEMOLYSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 6 (10) | 4 (4)
MYELOSUPPRESSION (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 33 (46) | 28 (31)
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3) | 5 (12)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 4 (5)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 1 (1)
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 9 (11)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 3 (3) | 2 (3)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 2 (2)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 2 (2)
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 (2) | 1 (1)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 5 (5)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 3 (3)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 3 (3)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
HEREDITARY MOTOR AND SENSORY NEUROPATHY (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
DEAFNESS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
CORNEAL OPACITY (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (6) | 10 (11)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0)
ASCITES (Gastrointestinal disorders) | 2 (2) | 1 (2)
COLITIS (Gastrointestinal disorders) | 2 (2) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 3 (3)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 7 (8) | 11 (12)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
FAECALOMA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROENTERITIS EOSINOPHILIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 4 (5)
INTESTINAL POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL VILLI ATROPHY (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1)
MIKULICZ'S SYNDROME (Gastrointestinal disorders) | 1 (2) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 5 (5)
OBSTRUCTIVE PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 4 (5)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 2 (2)
SUBACUTE PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
SWOLLEN TONGUE (Gastrointestinal disorders) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 9 (13) | 5 (5)
ADVERSE DRUG REACTION (General disorders) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 2 (2)
CHEST PAIN (General disorders) | 4 (4) | 1 (1)
CHILLS (General disorders) | 3 (3) | 4 (4)
CYST RUPTURE (General disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 1 (1) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (2) | 3 (3)
HYPERPLASIA (General disorders) | 0 (0) | 1 (1)
HYPERTHERMIA (General disorders) | 1 (1) | 0 (0)
ILL-DEFINED DISORDER (General disorders) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1)
INFUSION SITE EXTRAVASATION (General disorders) | 0 (0) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 3 (3) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 23 (24) | 37 (43)
STENT-GRAFT ENDOLEAK (General disorders) | 1 (1) | 0 (0)
SWELLING FACE (General disorders) | 1 (1) | 0 (0)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 1 (2)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 3 (3)
CHOLANGITIS (Hepatobiliary disorders) | 1 (2) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 6 (7) | 5 (6)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 2 (2)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1)
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 (0) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1)
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 (0) | 1 (1)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 0 (0) | 2 (2)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
HAEMOPHAGOCYTIC LYMPHOHISTIOCYTOSIS (Immune system disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 3 (3) | 0 (0)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 2 (2) | 0 (0)
ABDOMINAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS INTESTINAL (Infections and infestations) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 3 (3) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
ARTHRITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 3 (3) | 1 (1)
BACTERAEMIA (Infections and infestations) | 2 (2) | 1 (1)
BACTERIAL TRACHEITIS (Infections and infestations) | 0 (0) | 1 (1)
BK VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BREAST ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 3 (3) | 9 (9)
CAMPYLOBACTER INFECTION (Infections and infestations) | 0 (0) | 2 (2)
CATHETER SITE CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 3 (3) | 4 (4)
CHRONIC SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1)
COMPLICATED APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 2 (2)
DEVICE RELATED INFECTION (Infections and infestations) | 2 (2) | 1 (1)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
DISSEMINATED VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 2 (2) | 1 (2)
ENCEPHALITIS ENTEROVIRAL (Infections and infestations) | 0 (0) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0)
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
EPIGLOTTITIS (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 7 (7)
GASTROENTERITIS ESCHERICHIA COLI (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 9 (9) | 9 (9)
HERPES ZOSTER INFECTION NEUROLOGICAL (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER OTICUS (Infections and infestations) | 0 (0) | 1 (1)
INFECTED CYST (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 10 (11) | 6 (7)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 2 (2) | 3 (3)
INFLUENZA (Infections and infestations) | 0 (0) | 4 (4)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (9) | 13 (23)
MASTOIDITIS (Infections and infestations) | 1 (1) | 0 (0)
MENINGITIS ENTEROVIRAL (Infections and infestations) | 0 (0) | 1 (1)
MUCOSAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
NEUROBORRELIOSIS (Infections and infestations) | 1 (1) | 0 (0)
NEUTROPENIC INFECTION (Infections and infestations) | 1 (1) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 5 (8) | 6 (9)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
OESOPHAGEAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
OOPHORITIS (Infections and infestations) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1)
OTITIS MEDIA CHRONIC (Infections and infestations) | 0 (0) | 1 (1)
OVARIAN BACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PARAPHARYNGEAL SPACE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PELVIC ABSCESS (Infections and infestations) | 0 (0) | 2 (2)
PERIODONTITIS (Infections and infestations) | 0 (0) | 1 (1)
PERITONSILLAR ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECII INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 43 (51) | 51 (61)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 1 (1)
PNEUMONIA FUNGAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 2 (2)
Q FEVER (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (11) | 6 (7)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1)
RHINOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SCROTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 9 (9) | 14 (18)
SEPTIC SHOCK (Infections and infestations) | 2 (2) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (2) | 1 (1)
SINUSITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS FUNGAL (Infections and infestations) | 0 (0) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 2 (2) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
TUBO-OVARIAN ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 5 (7)
URINARY TRACT INFECTION (Infections and infestations) | 7 (7) | 8 (8)
UROSEPSIS (Infections and infestations) | 5 (6) | 4 (5)
VARICELLA ZOSTER SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 (1) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 4 (4) | 1 (1)
VIRAL MYOSITIS (Infections and infestations) | 0 (0) | 1 (1)
ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 19 (21) | 36 (42)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SEROMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 1 (1)
EASTERN COOPERATIVE ONCOLOGY GROUP PERFORMANCE STATUS WORSENED (Investigations) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 1 (1)
RESPIROVIRUS TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEITIS DEFORMANS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SERONEGATIVE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TEMPOROMANDIBULAR JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ACOUSTIC NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (4)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (7)
BENIGN LARYNGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER TRANSITIONAL CELL CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (6)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
DUCTAL ADENOCARCINOMA OF PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTRIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
GASTROINTESTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HODGKIN'S DISEASE NODULAR SCLEROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HODGKIN'S DISEASE STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HORMONE RECEPTOR POSITIVE BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
INTRAOCULAR MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LENTIGO MALIGNA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
NON-SMALL CELL LUNG CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SCHWANNOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SQUAMOUS CELL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
VULVOVAGINAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0)
BRACHIAL PLEXOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL HAEMATOMA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2) | 0 (0)
DEMENTIA (Nervous system disorders) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 3 (3) | 1 (1)
DIZZINESS POSTURAL (Nervous system disorders) | 0 (0) | 1 (1)
DYSDIADOCHOKINESIS (Nervous system disorders) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (1)
FACIAL PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
HYPERAMMONAEMIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
HYPOTONIA (Nervous system disorders) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 1 (1)
LETHARGY (Nervous system disorders) | 0 (0) | 2 (2)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
MONOPARESIS (Nervous system disorders) | 0 (0) | 1 (1)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0)
ORTHOSTATIC INTOLERANCE (Nervous system disorders) | 0 (0) | 1 (1)
ORTHOSTATIC TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 1 (2) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 3 (3) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 1 (2)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 3 (3) | 4 (4)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 5 (5)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
ABORTION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
DEVICE BREAKAGE (Product Issues) | 0 (0) | 1 (1)
ALCOHOL PROBLEM (Psychiatric disorders) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (2) | 3 (5)
EMOTIONAL DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 2 (2)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
SUBSTANCE-INDUCED PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 4 (4)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 1 (2) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 1 (1)
RENAL INFARCT (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL PAIN (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL PELVIS FISTULA (Renal and urinary disorders) | 0 (0) | 1 (1)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 1 (1)
OVARIAN MASS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PROSTATITIS (Reproductive system and breast disorders) | 2 (2) | 1 (1)
VAGINAL ULCERATION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VULVOVAGINAL PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE LUNG INJURY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (12)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PARANASAL CYST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PHARYNGEAL PARAESTHESIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (11)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS EXFOLIATIVE GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 1 (1)
EMBOLISM (Vascular disorders) | 3 (3) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 2 (3)
HYPERTENSIVE URGENCY (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 2 (2) | 7 (7)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab+Chemotherapy (N=692) | Obinutuzumab+Chemotherapy (N=698)
ANAEMIA (Blood and lymphatic system disorders) | 72 (95) | 75 (88)
LEUKOPENIA (Blood and lymphatic system disorders) | 91 (267) | 87 (222)
NEUTROPENIA (Blood and lymphatic system disorders) | 307 (777) | 348 (885)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 52 (79) | 90 (150)
ABDOMINAL PAIN (Gastrointestinal disorders) | 78 (95) | 69 (84)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 53 (60) | 57 (64)
CONSTIPATION (Gastrointestinal disorders) | 221 (301) | 249 (326)
DIARRHOEA (Gastrointestinal disorders) | 168 (253) | 207 (318)
DRY MOUTH (Gastrointestinal disorders) | 23 (25) | 36 (40)
DYSPEPSIA (Gastrointestinal disorders) | 50 (56) | 65 (82)
NAUSEA (Gastrointestinal disorders) | 338 (577) | 354 (594)
STOMATITIS (Gastrointestinal disorders) | 55 (71) | 54 (72)
VOMITING (Gastrointestinal disorders) | 151 (211) | 182 (242)
ASTHENIA (General disorders) | 44 (55) | 47 (56)
CHEST DISCOMFORT (General disorders) | 36 (43) | 43 (45)
CHILLS (General disorders) | 74 (99) | 126 (172)
FATIGUE (General disorders) | 277 (392) | 275 (390)
INFLUENZA LIKE ILLNESS (General disorders) | 35 (36) | 34 (38)
MUCOSAL INFLAMMATION (General disorders) | 44 (55) | 36 (41)
OEDEMA PERIPHERAL (General disorders) | 40 (47) | 46 (50)
PAIN (General disorders) | 35 (40) | 26 (28)
PYREXIA (General disorders) | 150 (231) | 200 (277)
BRONCHITIS (Infections and infestations) | 42 (53) | 47 (69)
CONJUNCTIVITIS (Infections and infestations) | 26 (30) | 35 (42)
HERPES ZOSTER (Infections and infestations) | 40 (46) | 70 (75)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 71 (105) | 59 (97)
NASOPHARYNGITIS (Infections and infestations) | 143 (224) | 135 (200)
ORAL HERPES (Infections and infestations) | 43 (48) | 46 (54)
PNEUMONIA (Infections and infestations) | 46 (59) | 47 (63)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 35 (43) | 39 (67)
RHINITIS (Infections and infestations) | 36 (49) | 59 (71)
SINUSITIS (Infections and infestations) | 47 (58) | 68 (92)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 132 (189) | 153 (217)
URINARY TRACT INFECTION (Infections and infestations) | 66 (100) | 75 (111)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 347 (569) | 416 (699)
WEIGHT DECREASED (Investigations) | 45 (49) | 35 (37)
DECREASED APPETITE (Metabolism and nutrition disorders) | 91 (103) | 98 (114)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 29 (43) | 48 (72)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 127 (160) | 144 (180)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 115 (143) | 99 (127)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 44 (56) | 40 (46)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 42 (49) | 40 (46)
MYALGIA (Musculoskeletal and connective tissue disorders) | 38 (43) | 53 (63)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 65 (79) | 66 (75)
DIZZINESS (Nervous system disorders) | 57 (69) | 75 (88)
DYSGEUSIA (Nervous system disorders) | 40 (44) | 38 (42)
HEADACHE (Nervous system disorders) | 123 (185) | 155 (229)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 49 (52) | 51 (62)
PARAESTHESIA (Nervous system disorders) | 51 (68) | 62 (71)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 47 (50) | 59 (68)
ANXIETY (Psychiatric disorders) | 29 (31) | 44 (47)
INSOMNIA (Psychiatric disorders) | 89 (98) | 113 (131)
COUGH (Respiratory, thoracic and mediastinal disorders) | 185 (248) | 221 (305)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 88 (101) | 112 (131)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 73 (87) | 82 (98)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 35 (41) | 42 (53)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 37 (40) | 27 (27)
ALOPECIA (Skin and subcutaneous tissue disorders) | 77 (78) | 90 (94)
DRY SKIN (Skin and subcutaneous tissue disorders) | 36 (39) | 40 (44)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 37 (43) | 37 (40)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 38 (46) | 32 (35)
PRURITUS (Skin and subcutaneous tissue disorders) | 94 (116) | 102 (124)
RASH (Skin and subcutaneous tissue disorders) | 131 (170) | 127 (162)
FLUSHING (Vascular disorders) | 40 (44) | 46 (56)
HOT FLUSH (Vascular disorders) | 25 (28) | 38 (43)
HYPERTENSION (Vascular disorders) | 50 (70) | 64 (100)
HYPOTENSION (Vascular disorders) | 28 (32) | 44 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT01332968/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT01332968/SAP_001.pdf